CLINICAL TRIAL: NCT01829997
Title: A Prospective, Post-Market Assessment Of NanOss Bioactive 3D in the Posterolateral Spine
Brief Title: Assessment of nanOss Bioactive 3D in the Posterolateral Spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pioneer Surgical Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NB3D012012
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-03

CONDITIONS: Degenerative Disc Disease; Spinal Stenosis; Spondylolisthesis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis; Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nanOss Bioactive 3D BVF (Experimental): Bilateral, instrumented posterolateral fusion surgery where nanOss Bioactive 3D will be hydrated with autologous BMA and placed bilaterally on a bed of local autograft bone spanning the transverse processes of the treated segment. If an interbody fusion is performed, only a PLIF or TLIF with PEEK IBF devices may be performed.
  Interventions: Device: nanOss Bioactive 3D BVF

INTERVENTIONS:
Device: nanOss Bioactive 3D BVF — nanOss Bioactive 3D BVF, combined with autograft and bone marrow aspirate, used in the posterolateral spine between L2 and S1. Instrumentation is required. Interbody fusion with PEEK device and autograft may or may not be performed.

SUMMARY:
Spine fusion is one of the most common procedures performed in spinal surgery. Several surgical techniques can achieve a solid union, but the intertransverse posterolateral fusion (PLF) is the most widely used. However, complications can develop when the bone graft material used is insufficient to achieve the desired fusion. With its unique properties, nanOss Bioactive 3D can be mixed with bone marrow aspirate (BMA) and autograft bone to obtain new bone growth during the healing process.

nanOss Bioactive 3D is approved for use in the U.S., however, additional information is useful to assess its efficacy in the posterolateral spine. The purpose of this study is to assess fusion results in the posterolateral spine using nanOss Bioactive 3D mixed with autograft bone and BMA. It is hypothesized that the use of nanOss Bioactive 3D will result in fusion at 12 months, with CT evidence of bridging trabecular bone, less than 3mm of translational motion, and less than 5 degrees of angular motion.

DETAILED DESCRIPTION:
The post market clinical investigation is designed to assess instrumented PLF using nanOss Bioactive 3D bone void filler with autograft bone and bone marrow aspirate in patients with symptomatic spinal stenosis secondary to degenerative disc disease (DDD) with up to Grade 1 spondylolisthesis at one or two adjacent levels from L2-S1 characterized by the inclusion and exclusion criteria.

Patients will be evaluated at Preop, discharge, 6 and 12 months. X-rays will be obtained at each visit; Additionally, a CT scan will be performed at the 12 month postoperative visit to assess fusion status.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age and skeletally mature.
* Symptomatic spinal stenosis secondary to DDD with up to Grade 1 spondylolisthesis at one or two adjacent levels from L2-S1 requiring instrumented PLF surgery.
* Completed a minimum of 6 months of non-operative treatment.
* Pre-operative objective evidence of primary diagnosis confirmed by appropriate imaging studies (AP, Lateral, Flexion and Extension images and an MRI or CT scan).
* Is willing and able to return for post-treatment exams according to the follow-up called for in the protocol.
* Is able to review, understand and sign the informed consent document.

Exclusion Criteria:

* Symptomatic at more than two levels.
* Has had previous fusion surgery at the level(s) to be treated (previous discectomy, laminotomy, laminectomy or nucleolysis at the level(s) to be treated < 6 months ago is ok).
* Has > 11 degrees lumbar scoliosis.
* Has > 40 BMI.
* Has > Grade 1 spondylolisthesis.
* Has osteoporosis (T-score of -2.5 or below), osteomalacia, Paget's disease or metabolic bone disease.
* Has a disease that significantly inhibits bone healing (e.g., diabetes type 1, renal failure, impaired calcium metabolism).
* Has a medical condition that requires or has a history of chronic steroid use (i.e., oral steroids), with the exception of inhaled/nasal corticosteroids steroids or has any medical condition that requires treatment with drugs known to interfere with bone healing.
* Has a neurological disease (e.g., Parkinson's disease), a psychosocial disorder (e.g., suicidal, diminished capacity) or has a history of substance abuse which would preclude accurate evaluation or limit the ability to comply with study requirements.
* Has either an active infection or infection at the site of surgery
* Has a systemic disease (e.g., AIDS, HIV, active hepatitis, tuberculosis)
* Has rheumatoid arthritis or other autoimmune disease.
* Has spinal tumors.
* Has an active malignancy (except non-melanoma skin cancer) or history of any invasive malignancy unless treated and in remission for at least five years.
* Has a known sensitivity or allergies to porcine collagen, PEEK, tantalum or titanium.
* Has active arachnoiditis.
* Has fractures of the epiphyseal plate or fractures for which stabilization of the fracture is not possible.
* Is a prisoner.
* Is involved in spinal litigation at the treated level(s).
* Is participating in another clinical study that would confound Study data.
* Is pregnant or is interested in becoming pregnant while participating in the Study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-04; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Robbins, MD, Principal Investigator — Milwaukee Spinal Specialists
Locations (4):
- United States (4):
  - Hospital for Joint Disease, New York, New York
  - Hospital for Special Surgery, New York, New York
  - MUSC Neurosurgery & Spine Services, Charleston, South Carolina
  - Milwaukee Spinal Specialists, Glendale, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | nanOss Bioactive 3D BVF
Started | 22
Completed | 16
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | nanOss Bioactive 3D BVF
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 60 [37 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Fusion
Description: Fusion is defined as the presence of bridging trabecular bone and less than 3mm of translational motion and less than 5mm of angular motion.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | nanOss Bioactive 3D BVF
Number analyzed (Participants) | 18
Participants | 16

2. Secondary Outcome: Number of Participants With Improvement in Quality of Life
Description: Number of participants with improvement in quality of life after surgery using the RAND-36 (a short form health survey). It is a 36 set of easily administered quality of life measures answered by the patient.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | nanOss Bioactive 3D BVF
Number analyzed (Participants) | 16
Participants | 16

3. Secondary Outcome: Number of Participants With Improvement in Pain Scores
Description: Number of participants with improvement in pain scores after surgery using the Visual Analog Scale. The scale measured from (0) no pain to (10) unbearable pain.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | nanOss Bioactive 3D BVF
Number analyzed (Participants) | 18
Participants | 18

4. Secondary Outcome: Number of Participants With Decreased Usage of Pain Medication
Description: Number of participants with decreased usage of pain medication after surgery
Time Frame: 12 months
Population: Data was not collected
Arm/Group | nanOss Bioactive 3D BVF
Number analyzed (Participants) | 0

5. Secondary Outcome: Returning to Work
Description: Time frame in which patient returned to work after surgery
Time Frame: 12 Months
Population: Data was not collected
Arm/Group | nanOss Bioactive 3D BVF
Number analyzed (Participants) | 0

6. Secondary Outcome: Satisfaction With Surgery
Description: Overall satisfaction with the procedure
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | nanOss Bioactive 3D BVF
Number analyzed (Participants) | 18
Participants | 18

ADVERSE EVENTS:
Time Frame: 2 years
Description: 0
Arm/Group | nanOss Bioactive 3D BVF
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 3/22
Other Adverse Events (participants affected / at risk) | 19/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | nanOss Bioactive 3D BVF (N=22)
Continued leg pain (Musculoskeletal and connective tissue disorders) | 1
Increased bilateral leg pain (Musculoskeletal and connective tissue disorders) | 1
Right iliac implant pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | nanOss Bioactive 3D BVF (N=22)
Right leg pain (Musculoskeletal and connective tissue disorders) | 7
Bilateral leg pain (Musculoskeletal and connective tissue disorders) | 2
Continued leg pain (Musculoskeletal and connective tissue disorders) | 1
Lower back pain (Musculoskeletal and connective tissue disorders) | 2
Hernia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Arm tingling (Musculoskeletal and connective tissue disorders) | 2
Bleeding hemorrhoids (General disorders) | 1
Altered mental status (General disorders) | 1
CSF Leak (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT01829997/Prot_SAP_000.pdf